CLINICAL TRIAL: NCT00380081
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study of the Efficacy and Safety of Sublingual Zolpidem Tartrate Tablet in Adult Patients With Insomnia Characterized by Difficulty Returning to Sleep After Middle-of-the-Night (MOTN) Awakening
Brief Title: A Study of Zolpidem Tartrate Sublingual Tablet in Adult Patients With Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Transcept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZI-06-010
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- placebo/zolpidem 3.5/zolpidem 1.75 (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet 3.5mg; Drug: zolpidem tartrate sublingual tablet 1.75mg; Drug: Placebo
- placebo/zolpidem 1.75/zolpidem 3.5 (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet 3.5mg; Drug: zolpidem tartrate sublingual tablet 1.75mg; Drug: Placebo
- zolpidem 3.5/placebo/zolpidem 1.75 (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet 3.5mg; Drug: zolpidem tartrate sublingual tablet 1.75mg; Drug: Placebo
- zolpidem 3.5/zolpidem 1.75/placebo (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet 3.5mg; Drug: zolpidem tartrate sublingual tablet 1.75mg; Drug: Placebo
- zolpidem 1.75/placebo/zolpidem 3.5 (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet 3.5mg; Drug: zolpidem tartrate sublingual tablet 1.75mg; Drug: Placebo
- zolpidem 1.75/zolpidem 3.5/placebo (Experimental)
  Interventions: Drug: zolpidem tartrate sublingual tablet 3.5mg; Drug: zolpidem tartrate sublingual tablet 1.75mg; Drug: Placebo

INTERVENTIONS:
Drug: zolpidem tartrate sublingual tablet 3.5mg — Zolpidem tartrate sublingual tablet 3.5 milligram administered between 2:15 and 3:15 a.m. on Night 1 and 2 of each treatment period. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.
  Other Names: Intermezzo®
Drug: zolpidem tartrate sublingual tablet 1.75mg — Zolpidem tartrate sublingual tablet 1.75 milligram administered between 2:15 and 3:15 a.m. on Night 1 and 2 of each treatment period. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.
  Other Names: Intermezzo®
Drug: Placebo — Placebo sublingual tablet administered between 2:15 and 3:15 a.m. on Night 1 and 2 of each treatment period. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.

SUMMARY:
The purpose of this study is to evaluate sleep onset following administration of Transcept zolpidem tartrate sublingual tablet versus placebo in adult insomnia patients.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia as defined by DSM-IV criteria and supported by subject diary
* Male or female between the ages of 18-64 years
* Body mass index (BMI) between 18-34 kg/m^2
* Females of childbearing potential must use a medically acceptable method of contraception
* Capable of understanding and willing to comply with study procedures and has provided informed consent

Exclusion Criteria:

* Females who are pregnant, breast-feeding or have a positive pregnancy test
* Any circadian rhythm disorder including planned travel across several time zones during the study period
* Known hypersensitivity to Zolpidem
* Has performed regular shift work with the past several months prior to screening
* An acute clinically significant illness or surgery as determined by the PI within 30 days of screening
* Patients that have used any central nervous system (CNS) medication or other medication known to impact the sleep/wake cycle
* A history of psychiatric disorder as defined by DSM-IV
* A history of drug addiction or alcohol abuse
* Any current significant disease, unless adequately controlled with a protocol allowed medication
* Known history of HIV or Hepatitis B or C
* Patients who have received an investigational drug within several months of screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roth, PhD, Principal Investigator — Henry Ford Hospital, Sleep Disorders and Research Center; Martin Scharf, PhD, Principal Investigator — Tri-State Sleep Disorders Center

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 83 patient volunteers were enrolled and of these, 82 patients were randomized, received at least 1 dose of study drug during the double-blind treatment period and were included in safety and efficacy analyses.
Groups:
- Placebo/Zolpidem 3.5/Zolpidem 1.75; Placebo/Zolpidem 1.75/Zolpidem 3.5; Zolpidem 3.5/Placebo/Zolpidem 1.75; Zolpidem 3.5/Zolpidem 1.75/Placebo; Zolpidem 1.75/Placebo/Zolpidem 3.5; Zolpidem 1.75/Zolpidem 3.5/Placebo: Cross-over interventions administered in the order listed.
Period: Overall Study
Arm/Group | Placebo/Zolpidem 3.5/Zolpidem 1.75 | Placebo/Zolpidem 1.75/Zolpidem 3.5 | Zolpidem 3.5/Placebo/Zolpidem 1.75 | Zolpidem 3.5/Zolpidem 1.75/Placebo | Zolpidem 1.75/Placebo/Zolpidem 3.5 | Zolpidem 1.75/Zolpidem 3.5/Placebo
Started | 14 | 13 | 13 | 15 | 13 | 14
Completed | 14 | 13 | 13 | 15 | 12 | 13
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Family Emergency | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Zolpidem 3.5/Zolpidem 1.75 | Placebo/Zolpidem 1.75/Zolpidem 3.5 | Zolpidem 3.5/Placebo/Zolpidem 1.75 | Zolpidem 3.5/Zolpidem 1.75/Placebo | Zolpidem 1.75/Placebo/Zolpidem 3.5 | Zolpidem 1.75/Zolpidem 3.5/Placebo | Total
Number analyzed (Participants) | 14 | 13 | 13 | 15 | 13 | 14 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 13 | 15 | 13 | 14 | 82
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.2 (10.21) | 47.2 (14.90) | 49.6 (10.74) | 45.0 (9.64) | 41.8 (13.33) | 43.5 (12.99) | 45.9 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 10 | 11 | 10 | 9 | 58
  Male | 6 | 3 | 3 | 4 | 3 | 5 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8 | 8 | 7 | 6 | 7 | 6 | 42
  Hispanic | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black | 5 | 5 | 4 | 9 | 6 | 7 | 36
  Asian/Pacific | 0 | 0 | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 13 | 15 | 13 | 14 | 82
Body Mass Index [Mean (Standard Deviation); unit: kilograms/square meters] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters | 27.72 (3.494) | 27.10 (4.164) | 27.27 (4.164) | 27.43 (3.717) | 25.92 (4.393) | 26.84 (2.681) | 27.06 (3.718)
Height [Mean (Standard Deviation); unit: centimeters] | 174.6 (9.353) | 166.4 (7.574) | 172.4 (10.740) | 167.2 (10.246) | 167.4 (8.775) | 169.8 (9.955) | 169.6 (9.700)
Number of Nights with Middle of the Night Awakening [Mean (Standard Deviation); unit: number of nights] — Number of nights with Middle of the Night (MOTN) Awakenings is based upon self-reports on more than or equal to 3 nights and completion of at least 7 days of the 10-day Screening Morning Sleep Diary.
  number of nights | 9.3 (0.99) | 9.4 (1.19) | 8.9 (1.38) | 9.3 (0.98) | 9.3 (1.11) | 8.6 (1.50) | 9.1 (1.20)
Weight [Mean (Standard Deviation); unit: kilograms] | 84.41 (11.409) | 75.10 (12.665) | 81.83 (17.816) | 77.46 (16.739) | 72.91 (14.421) | 77.50 (10.331) | 78.25 (14.249)

OUTCOME MEASURES:

1. Primary Outcome: Latency to Persistent Sleep After Middle-of-the-Night Awakening as Measured by Polysomnography
Description: Polysomnography was used to measure the time to return to persistent sleep after a middle-of-the-night (MOTN) awakening for each day of every two-day treatment period.
Time Frame: Days 1 and 2 for each treatment
Population: Intent-to-treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Groups:
- Zolpidem 3.5 mg: Zolpidem tartrate sublingual tablet 3.5 milligram administered between 2:15 and 3:15 a.m. on Night 1 and 2 of each treatment period. Participants placed the study drug under the tongue until it dissolved.
- Zolpidem 1.75 mg: Zolpidem tartrate sublingual tablet 1.75 milligram administered between 2:15 and 3:15 a.m. on Night 1 and 2 of each treatment period. Participants placed the study drug under the tongue until it dissolved.
- Placebo: Placebo sublingual tablet administered between 2:15 and 3:15 a.m. on Night 1 and 2 of each treatment period. Participants placed the study drug under the tongue until it dissolved.
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
minutes | 9.69 [8.06 to 11.65] | 16.89 [14.07 to 20.26] | 28.12 [23.41 to 33.77]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

2. Secondary Outcome: Number of Treatment Responders Based on Polysomnography Latency to Persistent Sleep After Middle-of-the-Night Awakening
Description: Polysomnography was used to measure the time to return to persistent sleep after a middle-of-the-night (MOTN) awakening for each day of every two-day treatment period. A participant was considered to be a responder if the time to return to persistent sleep was less than twenty minutes.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
participants | 60 | 46 | 23
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Treatment effect

3. Secondary Outcome: Total Sleep Time After Scheduled Middle-of-the-Night Awakening Measured by Polysomnography
Description: Polysomnography was used to measure the time from return to persistent sleep after a middle-of-the-night (MOTN) awakening until final awakening for each day of every two-day treatment period.
Time Frame: Days 1 and 2 for each treatment
Population: Intent-to-treat population.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
minutes | 208.99 [200.92 to 217.38] | 197.80 [190.23 to 205.68] | 183.12 [176.08 to 190.45]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

4. Other Pre Specified Outcome: Total Sleep Time After Scheduled Middle-of-the-Night Awakening Measured by Polysomnography for Participants With More Severe Insomnia
Description: Polysomnography was used to measure the time from return to persistent sleep after a middle-of-the-night (MOTN) awakening until final awakening for each day of every two-day treatment period in the subpopulation of patients with greater than 60 minutes to fall asleep after a MOTN awakening at baseline.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 37 | 38 | 37
minutes | 194.58 [179.72 to 210.65] | 179.98 [166.34 to 194.73] | 166.62 [153.90 to 180.39]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

5. Secondary Outcome: Average Subjective Total Sleep Time After Scheduled Middle-of-the-Night Awakening
Description: The time from return to persistent sleep after a middle-of-the-night (MOTN) awakening until final awakening for each day of every two-day treatment period was recorded by each participant using the Treatment Morning Sleep Questionnaire.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
minutes | 172.51 [161.92 to 183.10] | 162.36 [151.87 to 172.85] | 148.61 [138.07 to 159.15]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

6. Other Pre Specified Outcome: Latency to Persistent Sleep After Middle-of-the-Night Awakening as Measured by Polysomnography for a Subpopulation of Participants With More Severe Insomnia
Description: Polysomnography was used to measure the time to return to persistent sleep after a middle-of-the-night (MOTN) awakening for each day of every two-day treatment period in a subpopulation of patients with greater than 60 minutes to fall asleep after a MOTN awakening at baseline.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 37 | 38 | 37
minutes | 12.62 [9.12 to 17.47] | 23.28 [16.88 to 32.12] | 37.89 [27.38 to 52.43]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

7. Secondary Outcome: Subjective Sleep Quality Rating
Description: Sleep quality was rated by participants for each day of every two-day treatment period using the Treatment Morning Sleep Questionnaire. The percentage of participants within each rating category is reported. The rating scale was poor, fair, good and excellent.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
percentage of participants
  Poor | 18.8 | 29.3 | 34.6
  Fair | 38.8 | 37.8 | 42.0
  Good | 36.3 | 30.5 | 19.8
  Excellent | 6.3 | 2.4 | 3.7
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; The outcome noted above reflects the all-night sleep quality rating of study subjects who had a scheduled awakening after approximately 4 hours of sleep, were kept awake for 30 minutes and then allowed to return to bed and to sleep. After 4 hours, they were awakened again and disconnected from the PSG apparatus. Morning testing was conducted that included the Sleep Quality questionnaire. Evaluation of the results should reflect the nature of the study and the scheduled sleep disturbance; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Treatment effect

8. Secondary Outcome: Subjective Level of Refreshed Sleep
Description: Level of refreshed sleep was rated by participants for each day of every two-day treatment period using the Treatment Morning Sleep Questionnaire. The percentage of participants within each rating category is reported. The rating scale was poor, fair, good and excellent.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
percentage of participants
  Poor | 17.5 | 22.0 | 32.1
  Fair | 42.5 | 41.5 | 44.4
  Good | 35.0 | 34.1 | 19.8
  Excellent | 5.0 | 2.4 | 3.7
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.004, Cochran-Mantel-Haenszel — Treatment effect

9. Secondary Outcome: Subjective Ability to Function
Description: Ability to function was rated by participants for each day of every two-day treatment period using the Treatment Morning Sleep Questionnaire. The percentage of participants within each rating category is reported. The rating scale was poor, fair, good and excellent.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
percentage of participants
  Poor | 7.5 | 9.8 | 18.5
  Fair | 41.3 | 42.7 | 42.0
  Good | 45.0 | 41.5 | 33.3
  Excellent | 6.3 | 6.1 | 6.2
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel — Treatment effect

10. Secondary Outcome: Polysomnography Sleep Efficiency After Scheduled Middle-of-the-Night Awakening
Description: Sleep efficiency is a measurement of the percentage of time asleep to the total time in bed. It was measured by polysomnography for each day of every two-day treatment period.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time asleep
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
percentage of time asleep | 87.08 [83.73 to 90.57] | 82.63 [79.47 to 85.90] | 76.31 [73.38 to 79.35]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

11. Secondary Outcome: Subjective Sleep Onset Latency After Middle-of-the-Night Awakening
Description: Participants documented the time to return to sleep after a middle-of-the-night (MOTN) awakening for each day of every two-day treatment period using the Treatment Morning Sleep Questionnaire.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
minutes | 25.23 [21.58 to 29.49] | 28.58 [24.49 to 33.36] | 40.43 [34.62 to 47.23]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment effect

12. Secondary Outcome: Polysomnography Wake Time After Sleep Onset Following Middle-of-the-Night Awakening
Description: Amount of time awake after sleep onset following a middle-of-the-night awakening was measured by polysomnography for each day of every two-day treatment period.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
minutes | 15.06 [12.54 to 18.08] | 15.81 [13.18 to 18.97] | 15.71 [13.09 to 18.86]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p = 0.790, ANCOVA — Treatment effect

13. Secondary Outcome: Subjective Wake Time After Sleep Onset After Middle-of-the-Night Awakening
Description: Amount of time awake after sleep onset following a middle-of-the-night awakening was recorded by participants using the Treatment Morning Sleep Questionnaire for each day of every two-day treatment period.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 67 | 74 | 70
minutes | 28.69 [24.25 to 33.94] | 29.43 [25.03 to 34.62] | 34.22 [29.00 to 40.37]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p = 0.083, ANCOVA — Treatment effect

14. Secondary Outcome: Polysomnography Number of Awakenings After Middle-of-the-Night Awakening
Description: Number of times a participant awoke following sleep onset after the middle-of-the-night awakening, as measured by polysomnography for each day of every two-day treatment period.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: number of awakenings
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
number of awakenings | 3.71 [3.22 to 4.19] | 3.70 [3.22 to 4.18] | 4.13 [3.65 to 4.62]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p = 0.072, ANCOVA — Treatment effect
Statistical Analysis 2: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Period effect

15. Post Hoc Outcome: Subjective Number of Awakenings After Middle-of-the-Night Awakening
Description: Number of times a participant awoke following sleep onset after the middle-of-the-night awakening, as documented by the participant for each day of every two-day treatment period using the Treatment Morning Sleep Questionnaire.
Time Frame: Days 1 and 2 for each treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: number of awakenings
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Number analyzed (Participants) | 80 | 82 | 81
number of awakenings | 0.86 [0.70 to 1.04] | 1.03 [0.85 to 1.25] | 1.14 [0.94 to 1.39]
Statistical Analysis 1: Comparison: Zolpidem 3.5 mg vs Zolpidem 1.75 mg vs Placebo; Test type: Superiority or Other; p = 0.017, ANCOVA — Treatment effect

ADVERSE EVENTS:
Time Frame: Approximately one month
Arm/Group | Zolpidem 3.5 mg | Zolpidem 1.75 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/80 | 0/82 | 0/81

LIMITATIONS AND CAVEATS:
Scheduled nocturnal awakening is an established method used to evaluate treatments for naturally occurring middle-of-the-night awakenings. Additional studies are needed to determine the generalizability of the findings to 'real world' conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor agrees to review manuscripts within a reasonable period of time. If sponsor determines the publication included patentable subject matter, sponsor will be granted no less than 120 days to prepare patent applications.